CLINICAL TRIAL: NCT03569007
Title: A Phase 3, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Larazotide Acetate for the Relief of Persistent Symptoms in Patients With Celiac Disease on a GFD
Brief Title: Study to Evaluate the Efficacy and Safety of Larazotide Acetate for the Relief of CeD Symptoms
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial terminated by Sponsor
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CeD-LA-3001
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2021-08

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — larazotide acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Larazotide 0.25 mg (Active Comparator): Larazotide 0.25 mg capsules TID
  Interventions: Drug: Larazotide
- Larazotide 0.50 mg (Active Comparator): Larazotide 0.50 mg capsules TID
  Interventions: Drug: Larazotide
- Placebo (Placebo Comparator): Matching placebo capsules TID
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Larazotide — Synthetic 8-amino acid peptide formulated as enteric-coated beads in gelatin capsules
  Other Names: INN-202
  Arms: Larazotide 0.25 mg; Larazotide 0.50 mg
Drug: Matching Placebo — enteric-coated beads in gelatin capsules
  Other Names: placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of larazotide acetate versus placebo for the relief of persistent symptoms in adult celiac disease patients.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, placebo-controlled, multicenter, outpatient study to evaluate the efficacy and safety of larazotide acetate for the relief of persistent symptoms in adult patients with celiac disease on a gluten free diet.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults diagnosed with celiac disease (positive celiac serology plus confirmed biopsy) for at least 6 months
* On a gluten-free diet for at least 6 months
* Experiencing symptoms (ie, abdominal pain, abdominal cramping, bloating, gas, diarrhea, loose stool, or nausea)
* Willing to maintain current gluten-free diet throughout participation in the study

Exclusion Criteria:

* Refractory celiac disease or severe complications of celiac disease
* Chronic active GI disease other than celiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who are binary responders | 12 weeks
  Reduction in CeD PRO Abdominal Domain scores

CONTACTS AND LOCATIONS:
Locations (135):
- United States (135):
  - Research Site, Saraland, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, North Little Rock, Arkansas
  - Research Site, Bellflower, California
  - Research Site, Beverly Hills, California
  - Research Site, Canoga Park, California
  - Research Site, Corona, California
  - Research Site, Garden Grove, California
  - Research Site, Lancaster, California
  - Research Site, Los Gatos, California
  - Research Site, Northridge, California
  - Research Site, Poway, California
  - Research Site, Rialto, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Walnut Creek, California
  - Research Site, Bridgeport, Connecticut
  - Research Site, Bristol, Connecticut
  - Research Site, Hamden, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Inverness, Florida
  - Research Site, Lakewood Rch, Florida
  - Research Site, Miami, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Stone Mountain, Georgia
  - Research Site, Sugar Hill, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Idaho Falls, Idaho
  - Research Site, Arlington Heights, Illinois
  - Research Site, Fairview Heights, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Morton, Illinois
  - Research Site, Clive, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Crowley, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Catonsville, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Chesterfield, Michigan
  - Research Site, Rochester, Michigan
  - Research Site, Wyoming, Michigan
  - Research Site, Jackson, Minnesota
  - Research Site, Maplewood, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Petal, Mississippi
  - Research Site, Jefferson City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Freehold, New Jersey
  - Research Site, Ocean Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, Mineola, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Williamsville, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Concord, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Poland, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Happy Valley, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Scranton, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Warwick, Rhode Island
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, West Columbia, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, DeSoto, Texas
  - Research Site, Garland, Texas
  - Research Site, Harlingen, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Victoria, Texas
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Sandy City, Utah
  - Research Site, St. George, Utah
  - Research Site, Chesapeake, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Gainesville, Virginia
  - Research Site, Lansdowne Town Center, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Vancouver, Washington
  - Research Site, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No